CLINICAL TRIAL: NCT06852755
Title: Development of Biomarkers for Monitoring Menopause in Women
Status: Recruiting | Type: Observational
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FJUH112331
Record Dates: First submitted 2025-02-10; First posted 2025-02-28 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-02

CONDITIONS: Perimenopausal Biomarkers; Mitochondrial Biomarkers
Keywords: Perimenopausal Transition; Mitochondria; Biomarker; Women's Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — BLood, will use for checking female hormone (FSH, LH, estrogen, progesterone) and evaluate biomarker from the mitochondria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Reproductive Period: Women aged 20-40 years with regular menstrual cycles, representing the reproductive stage.
  Interventions: Other: Blood Sample Collection
- Perimenopausal Transition Period: Women aged 40-55 years have menstrual cycle within one year but experiencing menstrual irregularities, representing the transition into menopause.
  Interventions: Other: Blood Sample Collection
- Postmenopausal Period: Women aged 50 years and older who have not had a menstrual period for at least one year, representing the postmenopausal stage.
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Collection of peripheral blood samples for mitochondrial analysis, including the extraction of mononuclear cells and plasma for further assessment of mitochondrial quality and quantity.

SUMMARY:
This cross-sectional study aims to develop and validate mitochondrial biomarkers for monitoring menopause in women. The study will involve 100 participants divided into three groups: reproductive period, perimenopausal transition period, and postmenopausal period. Peripheral blood samples will be collected, and mitochondrial quality and quantity will be assessed using both qualitative and quantitative analyses. The study will identify potential biomarkers through metabolomics and validate them for monitoring the perimenopausal transition, providing a novel approach for women's health management during menopause.

DETAILED DESCRIPTION:
Background： Gender equality and equitable health have emerged as international trends in recent years. Despite existing solutions for women's health issues, many needs remain unmet. According to projections, the global menopausal population is expected to reach 1.2 billion by 2030, surpassing the prevalence of the most common chronic diseases. Presently, solutions exist for common menopausal symptoms such as hot flashes, night sweats, fatigue, irritability, and urinary incontinence. However, unresolved challenges encompass psychological changes and monitoring systems. Therefore, this project aims to develop biomarkers for menopause in women as a future monitoring system.

Most women enter menopause between the ages of 48 and 52. During this period, ovarian follicles cease activity, leading to the one-year period following the appearance of significant menstrual irregularities, known as the menopausal transition or perimenopause (1). As ovarian function gradually declines and estrogen secretion diminishes, various systemic changes occur, resulting in several menopause-related conditions such as osteoporosis, cardiovascular diseases, and urinary system issues. The decline in estrogen triggers a negative feedback loop, causing an increase in follicle-stimulating hormone (FSH) secretion and a reduction in E2 (17β-estradiol) production (2). Currently, menopausal hormone therapy (MHT) using estrogen can alleviate menopausal symptoms and restore overall E2 levels but doesn't lower FSH to premenopausal levels (3-4). However, a precise biomarker for monitoring menopause has not yet been established. Under estrogen deficiency, mitochondrial morphology and function may be compromised, while estrogen presence relates to reduced oxidative reactions, enhanced respiratory function, and stable membrane properties (5). This project aims to provide a comprehensive view through metabolomics to identify biomarkers within mitochondria that can be used for menopause monitoring.

Study Design： This study is a cross-sectional study. A total of 100 women will be included and grouped into three categories: 25 cases of reproductive period, 50 cases of perimenopausal transition period, and 25 cases of postmenopausal period. The peripheral blood will be collected. Following mitochondrial extraction, both qualitative and quantitative analyses are conducted. High-confidence protein markers are identified as candidate molecules using combined data from RNA-seq and LC/MS/MS. These candidate markers will undergo further validation testing.

Methods： After Ficoll separation, peripheral blood will be divided into mononuclear cells, plasma, and red blood cells. Further extraction of mitochondria will be carried out from both mononuclear cells and plasma. Quantitative experiments involve hippocampal measurements of metabolic energy and JC-1 assessment of mitochondrial health, while mitochondrial DNA copy number will be evaluated using digital PCR. Qualitative experimental analysis employs Western blotting to assess markers such as cytochrome c and HSP60 for mitochondria and PCNA for nuclear proteins. Candidate biomarker validation experiments use combined data from RNA-seq and LC/MS/MS to identify high-confidence protein markers as candidates, which are further validated for feasibility using the ELISA method.

Effect：

1. Understand the changes in mitochondrial quality and quantity during the perimenopausal transition in women.
2. Develop monitoring indicators for the perimenopausal transition in women.

ELIGIBILITY:
Inclusion Criteria:

* Biological female, age order than 20 years old.

Exclusion Criteria:

* Person with cancer.
* Person with any known acute or chronic infection.
* Person with known chronic illness under follow up or treatment.
* Pregnancy, one year withing delivery, under breast feeding, or three months within breast feeding.
* Under any female horemone therapy.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population Description: The study population consists of adult women aged over 20 years old, categorized into three groups:
  reproductive period (ages 20-45, regular menstrual cycles) perimenopausal transition period (ages 45-50, experiencing menstrual irregularities) postmenopausal period (ages over 50, no menstrual period for at least one year).
  All participants must be in general good health, without major chronic diseases, infection, or pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial Quantitative Analysis | 12 months from study start
  This outcome measure involves evaluating mitochondrial energy metabolism, including ATP content, oxygen consumption rate (OCR), and extracellular acidification rate (ECAR) using a hippocampal metabolic analyzer. Additionally, mitochondrial membrane potential will be assessed using flow cytometry to analyze the distribution of JC-1, indicating mitochondrial health. Digital PCR will be employed to measure mitochondrial DNA copy numbers, determining mitochondrial mass and comparing differences between groups.
Mitochondrial Qualitative Analysis | 12 months from study start
  This measure assesses mitochondrial protein markers using Western blot analysis. PCNA will be used as a nuclear protein marker, while cytochrome c and HSP60 will be used as mitochondrial protein markers to evaluate mitochondrial quality
Validation of Candidate Biomarkers | 12 months from study start
  This outcome measure focuses on the validation of high-confidence protein markers identified through RNA-Seq and LC-MS/MS data. The validation will be conducted using customized protein databases and further experiments to confirm the feasibility of these candidate biomarkers for monitoring perimenopausal transition.

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis SR, Lambrinoudaki I, Lumsden M, Mishra GD, Pal L, Rees M, Santoro N, Simoncini T. Menopause. Nat Rev Dis Primers. 2015 Apr 23;1:15004. doi: 10.1038/nrdp.2015.4. PMID 27188659
- [Background] Pellegrino A, Tiidus PM, Vandenboom R. Mechanisms of Estrogen Influence on Skeletal Muscle: Mass, Regeneration, and Mitochondrial Function. Sports Med. 2022 Dec;52(12):2853-2869. doi: 10.1007/s40279-022-01733-9. Epub 2022 Jul 30. PMID 35907119
- [Background] Karppinen JE, Tormakangas T, Kujala UM, Sipila S, Laukkanen J, Aukee P, Kovanen V, Laakkonen EK. Menopause modulates the circulating metabolome: evidence from a prospective cohort study. Eur J Prev Cardiol. 2022 Aug 5;29(10):1448-1459. doi: 10.1093/eurjpc/zwac060. PMID 35930503
- [Background] Powers MS, Schenkel L, Darley PE, Good WR, Balestra JC, Place VA. Pharmacokinetics and pharmacodynamics of transdermal dosage forms of 17 beta-estradiol: comparison with conventional oral estrogens used for hormone replacement. Am J Obstet Gynecol. 1985 Aug 15;152(8):1099-106. doi: 10.1016/0002-9378(85)90569-1. PMID 2992279